CLINICAL TRIAL: NCT01692340
Title: Novel 13C Carotenoids for Absorption and Metabolism Studies in Humans.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-09105; NCI-2011-03180 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: tomato; prostate cancer; metabolism
MeSH Terms: conditions — Prostatic Neoplasms | interventions — (all-E) phytoene; phytofluene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isotopically labeled lycopene (Experimental): We will administer 10 mg of isotopically labeled lycopene, phytoene or phytofluene mixed with olive oil and spread on an English muffin for consumption by participants.
  Interventions: Other: Isotopically labeled lycopene, phytoene or phytofluene
- Isotopically labeled phytoene (Experimental): We will administer 3.2 mg isotopically labeled lycopene, phytoene or phytofluene mixed with olive oil and spread on an English muffin for consumption by participants.
  Interventions: Other: Isotopically labeled lycopene, phytoene or phytofluene
- Isotopically labeled phytofluene (Experimental): We will administer 10 mg of isotopically labeled lycopene, phytoene or phytofluene mixed with olive oil and spread on an English muffin for consumption by participants.
  Interventions: Other: Isotopically labeled lycopene, phytoene or phytofluene

INTERVENTIONS:
Other: Isotopically labeled lycopene, phytoene or phytofluene — We will administer 10 mg of labeled carotenoid mixed with olive oil and spread on an English muffin for consumption by participants.

SUMMARY:
Tomatoes contain several compounds which may be beneficial for human health and prevention of disease, although this relationship is poorly understood and very controversial. This study uses a new technology to study the absorption and metabolism of three different compounds found in tomatoes. These compounds are called: phytoene, phytofluene, and lycopene. We hypothesize that by studying the absorption and metabolism of these compounds, we may be able to understand how the compounds may influence health and disease processes.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 21-70 years old.
* Body mass index of between 18 and 27 kg/m2 (inclusive).
* Eastern Cooperative Oncology Group (ECOG)performance status of O.
* Not currently be taking carotenoid supplements
* Have Blood Urea Nitrogen (BUN)/Creatinine (CR), liver enzymes, Complete Blood Count (CBC), and Prothrombin time (PT/PTT/INR) within normal limits.
* Have a hemoglobin level of at least 11 g /dL at the time of randomization.
* Voluntarily agree to participate and sign an informed consent document.

Exclusion Criteria:

* Have a known allergy or intolerance to tomatoes.
* Have a history of a nutrient malabsorption disease (such as celiac disease) or other metabolic disorders requiring special diet recommendations.
* Have uncontrolled hyperlipidemia (total cholesterol > 200 mg/dL, LDL > 160 mg/dL and serum triglycerides > 200 mg/dL) or lipidemia that may influence carotenoid pharmacokinetics or transport.
* Smoke tobacco products
* Have a history of pituitary hormone diseases that currently require supplemental hormonal administration (thyroid hormones, ACTH, growth hormone) or other endocrine disorders requiring hormone administration with the exception of diabetes and osteoporosis.
* Are taking certain medications (prescription or over-the-counter) such as Orlistat, which interfere with dietary fat absorption.
* Are taking complementary and alternative medications that at the discretion of the study physician Steven K. Clinton(SKC) may interfere with carotenoid absorption or metabolism.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Moran NE, Novotny JA, Cichon MJ, Riedl KM, Rogers RB, Grainger EM, Schwartz SJ, Erdman JW Jr, Clinton SK. Absorption and Distribution Kinetics of the 13C-Labeled Tomato Carotenoid Phytoene in Healthy Adults. J Nutr. 2016 Feb;146(2):368-76. doi: 10.3945/jn.115.220525. Epub 2015 Dec 16. PMID 26674763
- [Derived] Moran NE, Cichon MJ, Riedl KM, Grainger EM, Schwartz SJ, Novotny JA, Erdman JW Jr, Clinton SK. Compartmental and noncompartmental modeling of (1)(3)C-lycopene absorption, isomerization, and distribution kinetics in healthy adults. Am J Clin Nutr. 2015 Dec;102(6):1436-49. doi: 10.3945/ajcn.114.103143. Epub 2015 Nov 11. PMID 26561629
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We completed the first two arms of the study with isotopically labelled lycopene and phytoene, however our funding was exhausted after the second arm and we did not complete the isotopically labelled phytofluene arm.
Groups:
- Isotopically Labeled Lycopene: 10.2 mg of labeled carotenoid with a controlled meal.
  Consumption of an isotopically labeled carotenoid followed by pharmacokinetic studies for absorption and metabolism
- Isotopically Labeled Phytoene: 3.2 mg of labeled carotenoid with a controlled meal.
  Consumption of an isotopically labeled carotenoid followed by pharmacokinetic studies for absorption and metabolism
- Istotopically Labeled Phytofluene: 10 mg of labeled carotenoid with a controlled meal.
  Consumption of an isotopically labeled carotenoid followed by pharmacokinetic studies for absorption and metabolism
Period: Overall Study
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene | Istotopically Labeled Phytofluene
Started | 8 | 4 | 0
Completed | 8 | 4 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy subjects (6 males and 6 females) between the age of 21-33 yo (inclusive).
Groups:
- Isotopically Labeled Phytofluene: 10 mg of labeled carotenoid with a controlled meal.
  Consumption of an isotopically labeled carotenoid followed by pharmacokinetic studies for absorption and metabolism
- Total: Total of all reporting groups
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene | Isotopically Labeled Phytofluene | Total
Number analyzed (Participants) | 8 | 4 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 8 | 4 |  | 12
  >=65 years | 0 | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: years old] | 24 [21 to 31] | 27.7 [21.9 to 32.3] |  | 25.3 [21 to 32.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 |  | 6
  Male | 4 | 2 |  | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 1 | 1 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 7 | 3 |  | 10
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Plasma Half Life of Labeled Carotenoid
Description: We will study the half life of isotopically labeled carotenoids.
Time Frame: labelled lycopene: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose. Labelled phytoene: hourly for hours 0 - 15, then hours 17, 19 and 21 hours after dosing. Then, 1, 2, 3 4, 7, 10, 14, 17, 21 and 28 days post dose.
Measure: Mean (Standard Error); unit: days
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene
Number analyzed (Participants) | 8 | 4
days | 6.2 (0.3) | 2.3 (0.2)

2. Secondary Outcome: Carotenoid Metabolites
Description: Study the metabolites produced from the labeled carotenoid in healthy subjects
Time Frame: Up to 28 days
Population: Due to funding issues, at present we have not analyzed these samples for carotenoid metabolites. We have frozen plasma and if funds become available we would consider anlayzing the samples for carotenoid metabolites.
Groups:
- Isotopically Labeled Lycopene; Isotopically Labeled Phytoene: 10 mg of labeled carotenoid with a controlled meal.
  Consumption of an isotopically labeled carotenoid followed by pharmacokinetic studies for absorption and metabolism
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Maximal Plasma Carotenoid Concentration
Description: We will determine the average maximal plasma carotenoid concentration in healthy volunteers
Time Frame: 0 to 48 hours
Measure: Mean (Standard Error); unit: micromol
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene
Number analyzed (Participants) | 8 | 4
micromol | 0.14 (0.02) | 0.056 (0.006)

4. Primary Outcome: Time of Maximal Carotenoid Concentration
Description: We will determine when the maximal carotenoid concentration is achieved in the plasma
Time Frame: 0 to 48 hours
Measure: Mean (Standard Error); unit: hours
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene | Isotopically Labeled Phytofluene
Number analyzed (Participants) | 8 | 4 | 0
hours | 30 (6) | 19.8 (9.2) |

ADVERSE EVENTS:
Arm/Group | Isotopically Labeled Lycopene | Isotopically Labeled Phytoene
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes